CLINICAL TRIAL: NCT03066453
Title: Evaluation of an Antibiotic Treatment With 14 Days of Intravenous Tobramycin Versus the Same Antibiotic Associated With 5 Days of Intravenous Tobramycin Followed by Tobramycin Aerosol for 9 Days in Cystic Fibrosis.
Brief Title: Evaluation of Short Antibiotic Combination Courses Followed by Aerosols in Cystic Fibrosis
Acronym: TOBRAMUC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: new treatment that changes the management of the disease
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014_21; 2014-003882-10 (EudraCT Number); PHRC I 2013 (Other: number of funding)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis, tobramycin, antibiotic courses, FEV1
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard cure (Experimental): Antibiotic IV (Nebcin) 14 days and 14 days of tobramycin IV associated with one or more other antibiotic (s) IV in routine care
  Interventions: Drug: Tobi Inhalant Product; Drug: Nebcin
- Short cure (Experimental): antibiotic IV (Nebcin)14 days but with only 5 days of tobramycin IV followed 9 days of inhaled tobramycin (Tobi Inhalant Product) associated with one or more other antibiotic (s) IV in routine care
  Interventions: Drug: Tobi Inhalant Product; Drug: Nebcin

INTERVENTIONS:
Drug: Tobi Inhalant Product — inhaled tobramycin 300 mg twice per day
Drug: Nebcin — 10 to 12 mg/kg/day in 1 injection for adults and 10 to 15 mg/kg in 1 pediatric injection (combined with another IV antibiotic)

SUMMARY:
The aim of this study is to investigate the efficacy of antibiotic therapy with any antibiotic (IV) and IV (Nebcin®) tobramycin for 5 days followed by Solution for nebuliser inhalation (Tobi®) for 9 days and antibiotic cures using 14 days of tobramycin IV. In the case of positive results, the reduction of the duration of IV treatment of tobramycin from 14 days to 5 days would limit the risk of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis confirmed by sweat or genetic test
* Patient with clinical signs of exacerbation (increased cough, sputum (abundance, purulence), fever, anorexia, weight loss and FEV1) or acute exacerbations (defined at the clinician's discretion )
* FEV1 ≥ 25%
* Pseudomonas aeruginosa chronic carriers (defined by at least two antipyocyanic precipitation arcs or at least 3 successive positive ECBCs over a period of 18 months)
* Patient who received at least 1 IV course of antibiotics in the 18 months prior to inclusion.

Exclusion Criteria:

* Severe exacerbation (requiring hospitalization due to severe amputation of FEV 1, oxygen deficiency, or severe impairment of general health).
* Patient with 3rd antibiotic therapy (triple therapy)
* Patient colonized in Burkholderia cepacia
* Patient colonized by an atypical mycobacterium
* Patient with pulmonary transplant or transplant

  * chronic tinnitus
  * patient using hearing aid
* Hypersensitivity to tobramycin and other antibiotics of the aminoglycoside family
* Cirrhosis of Grades B and C according to the Child-Pugh Classification
* Myasthenia gravis
* Simultaneous administration of another aminoglycoside
* Renal failure
* Recent history of severe hemoptysis (within 2 months before inclusion)
* Patient participating simultaneously in another clinical study conducted on a drug for the duration of its participation in this research

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume at one second (FEV1) by spirometry | 18 months of the cure
  measure of dyspnea

SECONDARY OUTCOMES:
Forced expiratory volume at one second (FEV1) by spirometry | baseline and between day 16 or day 22
  measure of dyspnea
Visual Analog Scale | baseline and between day 16 or day 22
  measure of dyspnea, condition of patient, bronchial congestion
number of participants with Bronchial congestion | baseline and between day 16 or day 22
Sputum sample culture | baseline and between day 16 or day 22
  a descriptive analysis of Pseudomonas aeruginosa, and the other bacteria in the bacterial flora of sputum
Occurrence of the first exacerbation after the cure | during 18 months
Number of pulmonary exacerbations and those leading to hospitalization | during 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Prévotat, MD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - CRCM pédiatrique - CHU d'Amiens Hôpital Nord, Amiens
  - CRCM mixte - CHU de Caen Hôpital Côte de Nacre, Caen
  - CRCM mixte - CH de Dunkerque, Dunkirk
  - CRCM mixte - CH de Lens, Lens
  - CRCM adulte - CHRU de Lille Hôpital Calmette, Lille
  - CRCM pédiatrique - CHRU de Lille Hôpital Jeanne de Flandres, Lille
  - CRCM mixte - CHU de Rouen Hôpital Charles Nicolle, Rouen

IPD SHARING:
Plan to Share IPD: No